CLINICAL TRIAL: NCT03951779
Title: Diagnostic Utility of Exercise Cardiac Magnetic Resonance in the Assessment of Cardiac Dyspnea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Shapiro, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-005354
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Shortness of Breath; Cardiac; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with unexplained but suspected cardiac dyspnea (Experimental): Subjects with unexplained but suspected cardiac dyspnea who are being scheduled for right heart catheterization will undergo an exercise cardiac magnetic resonance imaging (eCMR).
  Interventions: Diagnostic Test: Exercise cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Exercise cardiac magnetic resonance imaging — Subjects will exercise on a treadmill and immediately following the completion of the stress protocol, subjects will undergo cardiac magnetic resonance imaging
  Other Names: eCMR

SUMMARY:
Researchers are examining the diagnostic utility of an exercise cardiac MRI (eCMR) in the assessment of cardiac dyspnea (shortness of breath).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged ≥18 years years with suspected cardiac dyspnea who are scheduled to undergo right heart catheterization as dictated by a comprehensive examination and echocardiography will be included for enrollment.

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Mechanical ventilation
* Acute or chronic renal failure (creatinine clearance <30 ml/min or requiring renal replacement therapy)
* Inability to perform MRI (i.e. claustrophobia, severe obesity (>150 kg), device incompatible with MRI)
* Inability to exercise
* Significant arrhythmia that precludes adequate ECG-gating for the MRI (i.e. atrial fibrillation with highly variable cycle lengths)
* Prior heart or lung transplantation
* Left ventricular systolic (ejection fraction <50%) or diastolic failure (based on Framingham criteria for heart failure with preserved ejection fraction)
* Significant left-sided valvular disease (≥moderate aortic stenosis, mitral stenosis, aortic regurgitation, mitral regurgitation) or prior valve surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Ejection Fraction | Baseline
  Measured using exercise cardiac magnetic resonance imaging (eCMR) reported in percentages
Stroke Volume | Baseline
  Measured using exercise cardiac magnetic resonance imaging (eCMG) reported in mL
Longitudinal Strain Assessment | Baseline
  Measured using exercise cardiac magnetic resonance imaging (eCMG) reported in percentages

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Shapiro, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials